CLINICAL TRIAL: NCT03122418
Title: Use of Personal Fitness Device in Adult (> 21 Years Old) Patients With Cystic Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 7754
Record Dates: First submitted 2017-04-17; First posted 2017-04-20 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Quality of Life

STUDY DESIGN:
Intervention Model Description: Subjects will receive a personal fitness device and asked to develop an individual exercise program.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise Study Group (Experimental): All subjects in this study will receive a personal fitness device and be asked to participate in some routine exercise. Each participant will be compared to their own initial CFQ-R score (to measure quality of life) before and after use of the personal fitness device.
  Interventions: Behavioral: Personal Fitness Device

INTERVENTIONS:
Behavioral: Personal Fitness Device — Subjects will be given a personal fitness device to use to encourage exercise routinely. The impact this has on the individual perception of their quality of life will be the primary outcome for this study

SUMMARY:
Approximately half of the variation in the presentation and disease status of patients with Cystic Fibrosis (CF) is secondary to non-genetic variables.[1] These include household income, compliance with therapy, second hand smoke exposure and possibly exercise (although exercise has less evidence to support its influence on disease status). Recently increased attention has been focused on the role of exercise and quality of life for patients with CF. This study will evaluate the role of exercise in relation to the patient's perception of their quality of life. The primary outcome will be the overall change in the patient's Cystic Fibrosis Questionnaire - Revised (CFQ-R) over a one year period during which the participants are encouraged to exercise and use a personal fitness device to track their exercise. This is a prospective single group non-blinded study. Participants will be asked to wear a personal fitness device for 11-13 months. The change in CFQ-R score is the primary outcome and other secondary outcomes will include; (1) exacerbations of cystic fibrosis (through use of antibiotics), (2) change in subject's FEV1, (3) inpatient admission rates, (4) change in BMI and (5) change in 6 minute walk test. The study will take place at the Adult CF Clinic on the University of Oklahoma Health Sciences Center campus.

DETAILED DESCRIPTION:
The specific aim of this study is to evaluate the use of personal fitness devices inpatients with cystic fibrosis over the age of 21.

The primary outcome will be the overall change in the patient's Cystic Fibrosis Questionnaire - Revised (CFQ-R) over a one year period. Secondary outcomes will evaluate (1) exacerbations of cystic fibrosis (through use of antibiotics), (2) change in subject's FEV1, (3) inpatient admission rates, (4) change in BMI and (5) change in 6 minute walk test

This is a prospective single group non-blinded study. Participants will be asked to wear a personal fitness device for 11-13 months (this will be the duration of their enrollment in the study). Upon enrollment, subjects will be given information regarding the benefits of physical activity and encouraged to develop an initial individual fitness goal. Two specific handouts regarding the benefits and how to start and exercise routine will be provided.

They will not be given a specific exercise program to follow, but instead will be encouraged to set personal fitness goals over the year and use the device to track these individual goals. Although they will be encouraged to have an individualized goal each participant will be asked to take a minimum of 5,000 steps per day during the first three months over the study and increase to 10,000 steps over the one year study period. This goal can be achieved by walking, aerobic classes or other exercise modalities, the method of exercise is expected to be variable for each participating subject and based on their personal preferences. Study participants individual goals will be noted by study staff during in the clinic visit in the electronic medical record. The personal fitness device to be used as part of this study is the Garmin Vivofit 2 fitness activity and sleep tracker.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosis of CF,
2. age of 21 or older,
3. willingness to consider some type of routine exercise,
4. BMI above 18 if female and above 20 for males,
5. willing to wear personal fitness device daily and
6. not already preforming daily exercise routinely

Exclusion Criteria:

1. patients who are unable or unwilling to understand and sign consent for this study,
2. patients who the study physicians determine it would not be safe to ask them to exercise,
3. patients who are not expected to survive over the next 12 months,
4. patients who are non-compliant and will not comply with study visits and procedures,
5. patients currently participating in other research trials,
6. patients who have had an acute exacerbation of their cystic fibrosis (treatment with oral or IV antibiotics) within the last 30 days,
7. patients with significant room air hypoxia who require more than 4 liters by nasal cannula to improve oxygenation to more than 90%.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2017-04-18 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Change in quality of life for individuals with CF using a personal fitness device | Will be completed upon enrollment and at 6 months and 12 months
  Will be measured using the CFQ-R questionnaire (a standard questionnaire for CF patients)

SECONDARY OUTCOMES:
Walking distance | This will be done upon enrollment, 6 months and 12 months
  Evaluate by a 6 minute walk test

CONTACTS AND LOCATIONS:
Overall Officials: Karen S Allen, MD, Principal Investigator — OUHSC
Locations (1):
- University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No
Initial data analysis was clear that study completion would not lead to a statistically significant difference in the primary outcome. Data are available and may be obtained through written request to the PI.